CLINICAL TRIAL: NCT04555746
Title: Children's Physical Activity Level and Sedentary Behaviour in Norwegian Early Childhood Education and Care: Effects of a Staff-led Cluster-randomized Controlled Trial
Brief Title: Active Kindergarten - Active Children
Acronym: AK-AC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Responsible Party: Principal Investigator, Eivind Andersen, Associate professor, University of South-Eastern Norway
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 1326
Record Dates: First submitted 2020-09-09; First posted 2020-09-21 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Healthy Lifestyle
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical activity (Experimental): Physical activity
  Interventions: Behavioral: Physical activity
- Control (No Intervention): Waiting list

INTERVENTIONS:
Behavioral: Physical activity — Four PA experts (researchers (PhD) within the field of PA and health in children, and physical education teachers) in collaboration with two members of the ECEC staff and two members of the municipality health department (paediatric physiotherapists) developed a frame for the intervention based on COP elements to be further developed, concretized and implemented by the staff. The intervention lasted for four months and contained the following components (Table 1): pre-meetings and follow up meetings in each ECEC institution; start up seminar and two follow up courses with all the staff members; ongoing planning and collective reflections practice in the ECEC institutions; Facebook group; and an equipment-package.
  Arms: Physical activity

SUMMARY:
The AK-AC study was designed as a two-arm, randomised by ECEC institution, evaluative controlled trial with the overarching aim of increasing the children's PA level and reduce sedentary time.

DETAILED DESCRIPTION:
Background A growing body of evidence suggests that children's physical activity (PA) level in childhood education and care (ECEC) settings is insufficient. Moreover, sedentary behaviour, defined as any waking behaviour characterized by an energy expenditure ≤ 1.5 metabolic equivalents while in a sitting, reclining, or lying posture, is highly prevalent and has been identified as detrimental to children's health. Although many children have healthy and active lifestyles, there seems to be a relatively large group of children with a low PA level. This could lead to negative developmental effects such as low fitness levels, weak motor skills and obesity. This is especially worrying because it is known that PA level often tracks from childhood into adulthood. Thus, early intervention is crucial given that PA plays a pivotal role in children's overall health and is associated with many positive health outcomes, including physical fitness, cardiovascular health, bone health and psychosocial and cognitive development.

PA levels have been found to be highly variable among children in ECEC settings and may therefore have great potential for effective interventions. Furthermore, since most children attend ECEC settings for many hours on most days of the week, and these institutions reach children across the socioeconomic spectrum, the ECEC setting may serve as an ideal avenue for increasing PA level, reducing sedentary time and enhancing the overall health of young children. However, early childhood educators identify parents rather than themselves as those responsible for promoting children's PA and may assume that young children receive adequate PA throughout the week regardless of their activities during their stay in the ECEC setting. Thus, intervening with children and staff in ECEC settings to equip them with the knowledge, abilities and motivation to promote PA in children during their ECEC time may provide substantial public health benefits.

In earlier studies, PA interventions conducted in ECEC settings have shown only small to moderate effects and were rather inconsistent across studies. Most PA interventions that have been implemented in ECEC settings have been structured programmes developed by PA experts and delivered by staff alone or with the strong influence of trained research personnel. In some studies, staff-led interventions have been shown to be less effective in increasing PA than interventions implemented by PA experts. Similar findings have emerged regarding intervention effects on fundamental movement skills. The main explanation for the lower efficiency of staff-led interventions may be that PA experts have more knowledge and competencies regarding this issue. For staff-led programmes to succeed, the need for multiple staff training sessions and maximizing the number of trained staff has been emphasized.

Recently, several reviews have summarized the body of knowledge regarding various aspects of the contexts of and prerequisites for PA in different kinds of out-of-home services for children of preschool age. A review including 34 studies revealed small but positive and significant intervention effects for children's (5 years) moderate- to vigorous-intensity PA (MVPA) but not for light-intensity PA. Based on their findings, the authors recommended interventions tailored to the target group and noted that cultural considerations, community needs and the provision of ongoing support should play key roles. Furthermore, they concluded that daily structured PA sessions, integrated into the everyday activities in the institutions (routines) and delivered through a hands-on approach, were most likely to contribute to increasing children's MVPA.

A review of 24 PA interventions in childcare, mostly targeting children between three and five years of age, where staff participated in professional development either before or during the intervention period and provided children with opportunities for additional PA. Less than half of the included studies had positive effects on children's PA level. For further intervention studies in ECEC, the authors provided four recommendations, of which two were based on the papers included in the review and two were based on evidence "from broader ECEC literature". First, there is a need for high-quality professional development prior to and during the intervention, and second, there is a need for "interventions that are 'outside the box'" in terms of, e.g., blended professional development; the role of technology; targeting the health, well-being and activity levels of the educators; focusing on PA learning experiences, outdoor time, and energy breaks; and integrating interventions into the institutions' daily routines. The third, broader-based recommendation addressed the importance of developing meaningful and trustworthy cooperation and relationships between staff and researchers. The fourth and final recommendation focused on the ECEC environment as a key factor for providing good opportunities for PA that thus should be increasingly emphasized in future interventions.

A missing perspective in recent studies focusing on PA interventions in ECEC settings might be that they do not fully take into account the fact that ECEC teaching professional practice has become increasingly complex due to increasingly diverse societies and multiple components related to working conditions. Thus, top-down approaches and standardized solutions (programmes) will possibly be difficult to implement in an ever more diverse environment in terms of individual, social, cultural and physical differences within and between institutions. Therefore, a suitable approach might be to establish organizational and collaborative learning processes, a community of professional learning, to improve and maintain staff competence. This means contextualizing pedagogical practice through continuous negotiation and reflection between staff members and through collective responsibility for improvement of practice instead of merely implementing structured programmes developed by external experts. While expert-delivered interventions seem to be best suited for effect studies, "real-world" approaches implemented by preschool teachers may have greater potential for developing sustainable and improved long-term practice.

The current study therefore suggests a dialogical and bottom-up approach that takes into account differences within and between local ECEC settings, such as child group characteristics; staff competencies, personal preferences and practices for sustainable implementation; differences in the physical indoor and outdoor environments; and available equipment to promote physically active play. Interventions that can be adapted to specific circumstances within an organization while maintaining overall fidelity are more likely to be successful. Hence, the theoretical frame of the current intervention is based on Wenger's theory on communities of practice (COP). Crucial for this theoretical perspective is the idea that organizations are learning communities that share competence and experiences to develop new practices. Such a community involves trusting in staff professionalism and their knowledge about and sensitivity towards the individual child and child groups as well as their awareness of barriers and possibilities in terms of environment and equipment. COP includes three modes of belonging: engagement, imagination and alignment. Engagement is actively participating in practice, revealing needs for learning and change and establishing the collective development of the organization. Imagination connects to the staff's visions and experience of meaning regarding the intervention, as well as their understanding of the purpose. Alignment is about commitment to the entire project. To achieve positive changes based on COP, these types of belonging must be linked to particular processes such as the establishment of mutual engagement over time to promote change, self-awareness and reflection on institutional practices. It is also important to transfer the knowledge and purpose of a practice across boundaries in the institution. A further key element is to establish practices where multiple perspectives are heard and appreciated to ensure that staff members can take advantage of opportunities to develop and experience themselves as acknowledged contributors to the institution. The current study, "Active Kindergarten - Active Children" (AK-AC), aims to examine the potential of a staff-led and expert-supported intervention to increase children's PA level and reduce sedentary time within the ECEC setting compared to standard care.

Methods Participants All children attending one of the 11 public ECEC institutions in Sandefjord municipality and born in 2011 (three- or four-year-olds) (n=130) were invited to participate in the study. Parents of a total of 116 children (89%) signed the informed consent form, and the children of these parents were included in the study. The intervention and control groups were formed at the centre level; six ECEC institutions were randomly assigned to the intervention group, and five institutions were assigned to the control group. The ECEC institutions varied in size and number of children (range 28 to 100 children). Most ECEC institutions follow the national recommended staff-child ratio of one staff member per three children under the age of three and per six children over the age of three. The regulations also demand one ECEC-educated teacher per nine children under the age of three and per 18 children over the age of three. The distribution showed a mixture of centre sizes in both the intervention and control group.

Intervention Four PA experts (researchers (PhD) within the field of PA and health in children and physical education teachers) in collaboration with two members of the ECEC staff and two members of the municipal health department (paediatric physiotherapists) developed a frame for the intervention based on COP elements to be further developed, concretized and implemented by the staff. The intervention lasted for four months and contained the following components: pre-meetings and follow-up meetings in each ECEC institution; a start-up seminar and two follow-up courses with all staff members; ongoing planning and collective reflection practice in the ECEC institutions; a Facebook group; and an equipment package.

ELIGIBILITY:
Inclusion Criteria:

* All children attending one of the 11 public ECEC institutions in Sandefjord municipality and born in 2011 (three or four year olds)

Exclusion Criteria:

* None

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Differences in accelerometer-measured physical activity and sedentary time at 4-month follow-up between intervention and control group | 5 days on both baseline and posttest
  Free-living PA was assessed using ActiGraph GT1M and GT3X+accelerometers (ActiGraph, LLC, Pensacola, FL, USA). The participants were instructed to wear the accelerometer on the left hip during their stay at the preschool for five consecutive days. The epoch length (sample interval) was set to 15 s. PA data were included if the participant had accumulated a minimum of 6 h of activity data per day for at least two days. The minutes spent in various levels of PA intensity were calculated. Sedentary behavior (sedentary time) was defined as ≤239 counts, light intensity PA was defined as 240 to 2119 counts, moderate intensity PA was defined as 2120 to 4449 counts, and any amount above 4450 was considered vigorous or very vigorous intensity PA.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen E, Ovreas S, Jorgensen KA, Borch-Jenssen J, Moser T. Children's physical activity level and sedentary behaviour in Norwegian early childhood education and care: effects of a staff-led cluster-randomised controlled trial. BMC Public Health. 2020 Nov 4;20(1):1651. doi: 10.1186/s12889-020-09725-y. PMID 33148218